CLINICAL TRIAL: NCT02283775
Title: A Phase 1b Study of SAR650984 (Isatuximab) in Combination With Pomalidomide and Dexamethasone for the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: SAR650984, Pomalidomide and Dexamethasone in Combination in RRMM Patients
Acronym: PomdeSAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD14079; U1111-1155-7484 (Other: UTN)
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PomdeSAR (Experimental): Part A: Isatuximab (escalating dose) on Day 1, 8, 15, and 22, then Day 1 and 15 + pomalidomide 4 mg on Day 1 to 21 + dexamethasone 40 mg (20 mg in patients of 75 years or older) on Day 1, 8, 15, 22 in 28-day cycles up to disease progression
  Part B: Isatuximab 10 mg/kg on Day 1, 8, 15, and 22, then Day 1 and 15 + pomalidomide 4 mg on Day 1 to 21 + dexamethasone 40 mg (20 mg in patients of 75 years or older) on Day 1, 8, 15, 22 in 28-day cycles up to disease progression
  Interventions: Drug: Isatuximab SAR650984; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form:solution for infusion Route of administration: intravenous
  Other Names: Sarclisa
Drug: Pomalidomide — Pharmaceutical form:capsules Route of administration: oral
  Other Names: Pomalyst
Drug: Dexamethasone — Pharmaceutical form:tablets or solution for infusion Route of administration: oral or intravenous

SUMMARY:
Primary Objectives:

Part A: To evaluate the safety and determine the recommended dose of SAR650984 in combination with pomalidomide (P) and dexamethasone (d), in patients with Relapsed/Refractory Multiple Myeloma (RRMM).

Part B: To evaluate the feasibility of isatuximab administered from a fixed infusion volume in combination with Pd as assessed by occurrence of grade ≥3 infusion associated reactions (IAR).

Secondary Objectives:

* To evaluate the infusion duration (Part B).
* To evaluate the safety profile of the combination with isatuximab administration from fixed volume (Part B).
* To evaluate immunogenicity of SAR650984 in combination with Pd (Part A and B).
* To evaluate the pharmacokinetics (PK) of SAR650984 and its effect on the PK of pomalidomide when administered in combination (Part A).
* To describe the efficacy of the combination of SAR650984 with Pd in terms of overall response rate and clinical benefit rate based on International Myeloma Working Group (IMWG) defined response criteria and the duration of response (Part A and B).
* To assess the relationship between clinical effects (adverse event [AE] and/or tumor response) and CD38 receptor density at baseline (Part A).

DETAILED DESCRIPTION:
The study duration for an individual patient will include a screening period for inclusion of up to 21 days. The treatment period may continue until disease progression, unacceptable adverse reaction, or other reason for discontinuation. After study treatment discontinuation an end of treatment (EOT) visit will be done at approximately 30 days after last study treatment component administration to assess safety. If the last ADA sample is positive or inconclusive, additional ADA will be sampled 3 months later. No further ADA will be sampled, even if this 3-month sample is positive. Patients who discontinue treatment for reasons other than progression of disease will be followed every month until progression or initiation of subsequent therapy, for a maximum of one year, whichever comes first.

ELIGIBILITY:
Inclusion criteria :

* Patient has been previously diagnosed with multiple myeloma (MM) based on standard criteria and currently requires treatment because MM has relapsed following a response, according to International Myeloma Working Group (IMWG) criteria.
* Patient had received at least two previous therapies including lenalidomide and proteasome inhibitor and have demonstrated disease progression on therapy or after completion of the last therapy.
* Patients with measurable disease defined as at least one of the following:

  * Serum M protein ≥0.5 g/dL (≥5 g/L);
  * Urine M protein ≥200 mg/24 hours;
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).

Exclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status >2.
* Poor bone marrow reserve.
* Poor organ function.
* Known intolerance/hypersensitivity to IMiDs, dexamethasone, boron or mannitol, sucrose, histidine or polysorbate 80.
* Any serious active disease (including clinically significant infection that is chronic, recurrent, or active) or co-morbid condition, which, in the opinion of the Investigator, could interfere with the safety, the compliance with the study or with the interpretation of the results.
* Any severe underlying medical conditions including presence of laboratory abnormalities, which could impair the ability to participate in the study or the interpretation of its results.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | Part A: Up to 4 weeks
Number of patients with adverse events and clinically significant changes in laboratory tests and vital signs according to the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) version 4.03 grade scaling | Part A: Up to 30 days for patients experiencing progressive disease and up to one year or the initiation of a new line of treatment for patients leaving the study for reasons other than progressive disease
Incidence of grade ≥3 IARs according to the NCI-CTC version 4.03 grade scaling | Part B: Up to 8 weeks

SECONDARY OUTCOMES:
Overall response rate | Part A: Up to approximately 8 months; Part B: Up to approximately 10 months
Pharmacokinetics: Partial area under the serum concentration time curve (AUC) | Part A: Up to approximately 10 months
Pharmacokinetics: maximum observed concentration (Cmax) | Part A: Up to approximately 10 months
Immune response: levels of human anti-human antibodies (ADA) | Part A: Up to approximately 8 months; Part B: Up to approximately 10 months
Duration of response - Time | Part A: Up to approximately 8 months; Part B: Up to approximately 10 months
Clinical Benefit rate | Part A: Up to approximately 8 months; Part B: Up to approximately 10 months
Infusion duration | Part B: Up to approximately 10 months
Safety of isatuximab administration from fixed volume | Part B: Up to 30 days for patients experiencing progressive disease and up to one year or the initiation of a new line of treatment for patients leaving the study for reasons other than progressive disease
Relationship between clinical effect and CD38 receptor density | Part A: Up to approximately 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (13):
  - Investigational Site Number 840001, Scottsdale, Arizona
  - Investigational Site Number 840006, Duarte, California
  - Investigational Site Number 840018, New Haven, Connecticut
  - Investigational Site Number 840011, Decatur, Illinois
  - Investigational Site Number 840004, Boston, Massachusetts
  - Investigational Site Number 840104, Boston, Massachusetts
  - Investigational Site Number 840010, Chapel Hill, North Carolina
  - Investigational Site Number 840003, Charlotte, North Carolina
  - Investigational Site Number 840014, Canton, Ohio
  - Investigational Site Number 840016, Charleston, South Carolina
  - Investigational Site Number 840015, Salt Lake City, Utah
  - Investigational Site Number 840005, Seattle, Washington
  - Investigational Site Number 840017, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Usmani SZ, Karanes C, Bensinger WI, D'Souza A, Raje N, Tuchman SA, Sborov D, Laubach JP, Bianchi G, Kanagavel D, Saleem R, Dubin F, Campana F, Richardson PG. Final results of a phase 1b study of isatuximab short-duration fixed-volume infusion combination therapy for relapsed/refractory multiple myeloma. Leukemia. 2021 Dec;35(12):3526-3533. doi: 10.1038/s41375-021-01262-w. Epub 2021 May 28. PMID 34050260
- [Derived] Mikhael J, Belhadj-Merzoug K, Hulin C, Vincent L, Moreau P, Gasparetto C, Pour L, Spicka I, Vij R, Zonder J, Atanackovic D, Gabrail N, Martin TG, Perrot A, Bensfia S, Weng Q, Brillac C, Semiond D, Mace S, Corzo KP, Leleu X. A phase 2 study of isatuximab monotherapy in patients with multiple myeloma who are refractory to daratumumab. Blood Cancer J. 2021 May 12;11(5):89. doi: 10.1038/s41408-021-00478-4. No abstract available. PMID 33980831
- [Derived] Mikhael J, Richardson P, Usmani SZ, Raje N, Bensinger W, Karanes C, Campana F, Kanagavel D, Dubin F, Liu Q, Semiond D, Anderson K. A phase 1b study of isatuximab plus pomalidomide/dexamethasone in relapsed/refractory multiple myeloma. Blood. 2019 Jul 11;134(2):123-133. doi: 10.1182/blood-2019-02-895193. Epub 2019 Mar 12. PMID 30862646